CLINICAL TRIAL: NCT00291265
Title: Testing Objective Measures of Motor Impairment in Early Parkinson's Disease
Brief Title: Measures of Motor Impairment in Early Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060096; 06-N-0096
Record Dates: First submitted 2006-02-11; First posted 2006-02-13 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-02-02

CONDITIONS: Parkinson's Disease
Keywords: Bradykinesia; Tremor; Speech; Rigidity; Neurodegeneration; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease; Hypokinesia; Tremor; Speech; Muscle Rigidity; Nerve Degeneration

SUMMARY:
This study will test the accuracy of a new home-use electronic device that measures and records small changes in Parkinson's disease symptoms, such as tremor and impaired movement and speech. The testing is done at home and the results are sent by Internet to the patient's doctor. Detecting Parkinson's disease in its early stages may permit doctors to provide early treatment and slow the rate of disease progression.

Patients with early Parkinson's disease (less than 5 years) with rest tremors and bradykinesia (slowness and difficulty of movement) who are not taking medications for the disease may be eligible for this study. Candidates are screened with training and practice in using the home monitoring device over 2-3 weeks. Those who demonstrate proficiency with the device may be enrolled in the study.

Participants undergo the following tests and procedures:

Baseline Visit

Participants' undergo symptoms ratings using the Unified Parkinson's Disease Rating Scale and assessments of memory, thinking and depression.

At-home testing

Participants begin at-home testing with the monitoring device after the baseline visit and repeat the tests weekly for 6 months. The test information is automatically uploaded to a home computer (provided by the study) and sent to the investigators via Internet. The test procedure is as follows:

* Introduction questionnaire (1 minute): Participants are questioned about how they are feeling at test time.
* Pegboard test (4 minutes): At the sound of a tone, the participant moves eight pegs from the right to the left using their right and then left hand.
* Tapping test (3 minutes): At the sound of a tone, the participant alternately presses two buttons with the right index finger and then the left index finger.
* Reaction time/movement time testing (3 minutes): At the sound of a tone, the participant moves his or her index finger from one button to the other, first with the right hand and then with the left hand.
* Digitography testing (4 minutes): At the sound of a tone, the participant alternates between pressing two keys with the index and middle fingers.
* Speech + Actiwatch tremor data upload (7 minutes): The participant: 1) takes a deep breath and says "ahhh" for as long as possible; 2) is shown a picture and, at the sound of a tone, is asked to tell a story about the picture; 3) uploads the tremor data from the Actiwatch (a device worn on the wrist that records tremors).
* At specified times du...

DETAILED DESCRIPTION:
Objective: Because neuroprotective strategies in Parkinson's disease are primarily aimed at intervening in the early phase of disease, appropriate measures of minor, subtle parkinsonian impairments need to be defined. The gold standard of rating scales for Parkinson's disease is the Unified Parkinson's Disease Rating scale (UPDRS), but it covers the gamut of disability levels and does not specifically focus on early impairments. We have developed a series of motor tasks that can be performed with a home-based computer module so that data can be collected frequently and prospectively without obligating the patient to come to a medical center.

Study population: The study population will consist of patients with mild and early Parkinson disease.

Design: This feasibility study will longitudinally follow 50 patients with mild and early Parkinson's disease who are not receiving symptomatic therapy for the treatment of motor impairment. They will be trained to perform the task and transmit data on a weekly basis.

Outcome measures: We will analyze time-related changes in several domains of motor function (tremor, limb bradykinesia, fine motor bradykinesia, voice, reaction time/movement time) and correlate these changes with the UPDRS at 3 and 6 months. We hypothesize that patients will find this assessment technology easy to use, a positive force in their lives, and that they will be committed to the program throughout its duration. Further, we hypothesize that motor changes will be detected with this technology at a time when UPDRS scores do not show decrements. Over six months, however, declines in the UPDRS will occur and correlate with the decrements in computer-based motor task. If, as we hypothesize, the home-based motor testing program is both feasible and useful in the assessment of early impairments in Parkinson's disease, it will be particularly applicable to neuroprotective trials currently being designed.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. PD, defined with at least two of the following cardinal features: rest tremor, bradykinesia, rigidity with PD diagnosis less than or equal to 5 years.
  2. Hoehn and Yahr stage less than 3.
  3. No clinical evidence of other parkinsonian syndromes (Progressive supranuclear palsy, Multiple system atrophy, drug-induced parkinsonism, lewy body dementia).
  4. The patient must not be on any drug therapy for symptomatic control of parkinsonism, specifically levodopa, dopamine agonist, amantadine, anticholinergic drugs, COMT-inhibitors, selegiline while participating in the initial 6 months of the study.
  5. Patients must express a willingness and intent to remain off all medications that could affect parkinsonism for the first 6 months of the study without first informing the site PI. Starting an anti-Parkinson medication does not necessarily disqualify a patient from continuing with the study. After the initial 6 months of participation, the patients will be allowed to start a anti-Parkinson medications.
  6. Patient must express a willingness and intent to remain off of all medications that could affect parkinsonism for the first 6 months of the study without first informing the site PI. Starting an anti-Parkinson medication does not necessarily disqualify a patient from continuing with the study. After the initial 6 months of participation, the patients will be allowed to start anti-Parkinson medications.
  7. Patient must demonstrate proficiency in the use of the At Home Testing Program in an office setting.
  8. Participants must be willing to have a technician come to their homes to set up the equipment, check on it periodically, and remove it at study end.

EXCLUSION CRITERIA:

1. Patients who have comorbid neurological or psychiatric disorders (even if they don't require medications).
2. Patients who have had Parkinson's disease for more than 5 years.
3. Patients who have another movement disorder (Progressive supranuclear palsy, Multiple system atrophy, drug-induced parkinsonism, Lewy body dementia).
4. Disruptive non-compliance with requirements of the study causing an inability to collect valid and clean data.
5. Inability to accurately perform the task required of this study (i.e. cannot use the equipment properly and to transfer data using a simple USB connection).

Please note that there is no inclusion or exclusion criteria based on depression or dementia. However, if these problems interfered with proficiency of data acquisition during the screening phase, they will not be eligible. The Hamilton Depression Rating Scale will be the measure used. Depression scale scores will be used as potential co-variants to compliance in exploratory analysis. Furthermore, treatment of other medical conditions will be allowed during the treatment period. Treatment of any feature of Parkinson's disease that does not involve the exclusionary medications (see inclusion/exclusion criteria) will be allowed.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-02-09; Study Completion 2010-02-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Adler CH, Hentz JG, Joyce JN, Beach T, Caviness JN. Motor impairment in normal aging, clinically possible Parkinson's disease, and clinically probable Parkinson's disease: longitudinal evaluation of a cohort of prospective brain donors. Parkinsonism Relat Disord. 2002 Dec;9(2):103-10. doi: 10.1016/s1353-8020(02)00012-3. PMID 12473400
- [Background] Bloem BR, Beckley DJ, van Hilten BJ, Roos RA. Clinimetrics of postural instability in Parkinson's disease. J Neurol. 1998 Oct;245(10):669-73. doi: 10.1007/s004150050265. PMID 9776467
- [Background] Bronte-Stewart HM, Ding L, Alexander C, Zhou Y, Moore GP. Quantitative digitography (QDG): a sensitive measure of digital motor control in idiopathic Parkinson's disease. Mov Disord. 2000 Jan;15(1):36-47. doi: 10.1002/1531-8257(200001)15:13.0.co;2-m. PMID 10634240